CLINICAL TRIAL: NCT01232699
Title: Internet Obesity Treatment Enhanced With Motivational Interviewing
Acronym: iReach2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Principal Investigator, Jean R. Harvey, PhD, RD, Principal Investigator, University of Vermont
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-124
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Obesity
Keywords: obesity; weight loss; internet treatment; motivational interviewing
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Internet Obesity Treatment (Active Comparator): Participants will attend weekly class sessions on line and track food and exercise in an on-line journal.
  Interventions: Behavioral: Internet Obesity Treatment
- Internet Obesity Treatment with MI (Experimental): Participants will attend weekly classes on line, record food and exercise in an on-line journal, and will have no more than 6 individual motivational interviewing sessions.
  Interventions: Behavioral: Internet Obesity Treatment with MI
- Contingent MI (Experimental): Intervention is the same as for the MI arm, however participants will only receive MI if meeting certain treatment participation conditions.
  Interventions: Behavioral: Contingent MI

INTERVENTIONS:
Behavioral: Internet Obesity Treatment — Participants will engage in self monitoring, will receive skills training to help cope with environmental triggers, and will receive nutrition advice.
  Other Names: iREACH2
  Arms: Internet Obesity Treatment
Behavioral: Internet Obesity Treatment with MI — In addition to weekly group meetings, self-monitoring through recording calorie and fat intake daily as well as exercise, participants will meet one-on-one with an MI counselor on-line in order to augment an individual's motivation to change behavior.
  Other Names: iREACH2
  Arms: Internet Obesity Treatment with MI
Behavioral: Contingent MI — Participants will attend weekly behavioral internet meetings. They may or may not receive Motivational Interviewing depending on their class attendance.
  Other Names: iReach2
  Arms: Contingent MI

SUMMARY:
Internet-based weight control programs have been shown effective in producing weight loss, but in-person delivery of behavioral weight control produces significantly greater weight loss than on-line delivery of the same program. Motivational Interviewing has been shown to increase weight loss when delivered as an adjunct to in-person weight loss programs but has not been examined in conjunction with web-based obesity treatment. Therefore, the overall goal of this project is to determine if the addition of on-line Motivational Interviewing to a web-based group behavioral obesity treatment program will augment weight loss outcomes.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to determine whether weight losses in a group behavioral weight loss intervention conducted over the Internet are increased with the inclusion of individual, online MI sessions. All participants will receive the same online 6-month group-based behavioral weight loss program followed by 12 months of weight maintenance. Overweight and obese adults at two study sties (N=426) will be randomized to (1) Internet intervention; or 2) Internet intervention with individual MI sessions occurring at three month intervals on a fixed schedule (Internet+MI-Fixed). Assessments will be conducted every six months and will include measures of body weight and height, diet and exercise behaviors, Quality of Life, adherence measures (eg., attendance, compliance with self-monitoring), social influence components, motivation, treatment satisfaction, demographic data and descriptive information regarding use of website components. A third arm was added for the final 3 intervention cohorts. All participants received the program as described above with the addition of motivational interviewing contingent on participants' attendance in classes.

ELIGIBILITY:
Inclusion Criteria:

* must be over 18
* must have a BMI between 18 and 50
* must live within 60 minutes driving distance of University of Arkansas, Little Rock, AR, or University of Vermont, Burlington, Vermont
* must be able to walk for exercise

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2010-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | 6 months
  Weights will be taken in street clothes without shoes using a hospital quality digital floor model scale.
Change in Body Weight | 12 months
Change in Body Weight | 18 months
Change in body weight | 0
  Weights will be taken in street clothes without shoes using a hospital quality digital floor model scale. Height will be taken at baseline using a wall-mounted stadiometer and BMI will be calculated as weight (kg)/height(m2)

SECONDARY OUTCOMES:
Adherence to Treatment Components | 6 months
  Items will include attendance at chat group meetings and completion of online food diaries and exercise records.
Adherence to Treatment Components | 12 months
Adherence to Treatment Components | 18 months
Motivation Measures | 0
  We will assess participant motivation for participating in a weight reduction program and adhering to the program.
Motivation Measures | 6
Motivation Measures | 12 months
Motivation Measures | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean R Harvey Berino, PhD., Principal Investigator — University of Vermont; Delia Smith-West, PhD., Principal Investigator — UAMS
Locations (2):
- United States (2):
  - University of Arkansas for the Medical Sciences, Little Rock, Arkansas
  - Behavioral Weight Management Program/Univ of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Harvey J, Krukowski R, Priest J, West D. Log Often, Lose More: Electronic Dietary Self-Monitoring for Weight Loss. Obesity (Silver Spring). 2019 Mar;27(3):380-384. doi: 10.1002/oby.22382. PMID 30801989
- [Derived] West DS, Harvey JR, Krukowski RA, Prewitt TE, Priest J, Ashikaga T. Do individual, online motivational interviewing chat sessions enhance weight loss in a group-based, online weight control program? Obesity (Silver Spring). 2016 Nov;24(11):2334-2340. doi: 10.1002/oby.21645. Epub 2016 Sep 12. PMID 27616628
- [Derived] Krukowski RA, DiLillo V, Ingle K, Harvey JR, West DS. Design and Methods of a Synchronous Online Motivational Interviewing Intervention for Weight Management. JMIR Res Protoc. 2016 Apr 19;5(2):e69. doi: 10.2196/resprot.5382. PMID 27095604